CLINICAL TRIAL: NCT07200206
Title: A Prospective, Single-arm, Non-interventional, Multi-center, Post-marketing Surveillance Study of Beyfortus (Nirsevimab) in Republic of Korea
Brief Title: A Post-marketing Surveillance Study of Beyfortus (Nirsevimab) in Republic of Korea
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: VAS00011; U1111-1316-0081 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-09-29; First posted 2025-10-01 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Syncytial Virus
MeSH Terms: interventions — nirsevimab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Children up to 24 months of age who are scheduled to receive Beyfortus according to the approved indications will be selected as participants under the real-world clinical practice settings during the surveillance period.
  Interventions: Biological: Nirsevimab

INTERVENTIONS:
Biological: Nirsevimab — Route of Administration: Intramuscular Pharmaceutical Form: Solution for injection
  Other Names: Beyfortus™

SUMMARY:
This study is conducted as part of the local risk management plan to collect and understand the following information about the surveillance drug under the real-world clinical practice settings.

To evaluate the safety of Beyfortus in Korean children who received Beyfortus under the real-world clinical practice settings per the approved indication. The investigator will decide whether to enroll participants if they determine that administering Beyfortus according to current practice can provide clinical benefits in terms of safety and efficacy Participants will be followed-up for 180 days after Beyfortus administration.

ELIGIBILITY:
Inclusion Criteria:

* Children up to 24 months of age who received Beyfortus according to the approved indications.
* Informed consent signed by the parents / legally accepted representatives (LARs) of the participant.

Exclusion Criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding the enrollment) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device or a medical procedure.
* Any contraindications according to the approved local product label of Beyfortus.

Ages: 0 Days to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children up to 24 months of age who are scheduled to receive Beyfortus according to the approved indications will be selected as participants under the real-world clinical practice settings during the surveillance period after the contract date at the institution. The participants must meet all study inclusion criteria and must not meet any of the study exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2029-09-26 (Estimated); Study Completion 2029-09-26 (Estimated)

PRIMARY OUTCOMES:
Occurence of Adverse Events (AEs) | Up to 180 days post dose
  Number of participants (and occurrences) experiencing AEs will be assessed.
Occurence of Serious Adverse Events (SAEs) | Up to 180 days post dose
  Number of participants (and occurrences) experiencing SAEs will be assessed.
Occurrence of AE of special interest (AESI) | Up to 180 days post dose
  Number of participants (and occurrences) experiencing AESI will be assessed. The definition of AESI is as follow:
  1. Hypersensitivity, including anaphylaxis
  2. Immune complex disease
  3. Thrombocytopenia
Occurence of Adverse Drug Reaction (ADRs) as Specified in Approved Local Label | Up to 180 days post dose
  Number of participants (and occurrences) experiencing ADRs will be assessed.
Occurrence of Respiratory Syncytial Virus (RSV) Lower Respiratory Tract Infection (LRTI) | Up to 180 days post dose
  Number of participants (and occurrences) experiencing RSV LRTI will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Nam Seung Woo Pediatric: 4100007, Hwaseong-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org